CLINICAL TRIAL: NCT00625937
Title: A Phase ll Trial of Induction Docetaxel and S-1 Followed by Concomitant Radiotherapy With Low-dose Daily Cisplatin in Locally Advanced Head and Neck Cancer
Brief Title: Docetaxel and S-1 Followed By Radiation Therapy and Low-Dose Cisplatin in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000582621; YONSEI-4-2006-021-0
Record Dates: First submitted 2008-02-28; First posted 2008-02-29 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cisplatin; Docetaxel; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Drug: tegafur-gimeracil-oteracil potassium
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, S-1, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving more than one drug (combination chemotherapy) together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel and S-1 together with radiation therapy and low-dose cisplatin works in treating patients with stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the response rate in patients with stage III or IV head and neck cancer treated with induction therapy comprising docetaxel and S-1 followed by radiotherapy and low-dose cisplatin.

Secondary

* To assess the effect of this regimen on survival and locoregional and systemic control rates in these patients.

OUTLINE:

* Induction chemotherapy: Patients receive oral S-1 twice daily on days 1-14 and docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
* Chemoradiotherapy: Patients receive low-dose cisplatin IV once daily and undergo radiotherapy 5 days a week for 7 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed head and neck cancer arising from the oral cavity, oropharynx, hypopharynx, or nasopharynx, including any of the following subtypes:

  * Squamous cell carcinoma
  * Poorly differentiated carcinoma
  * Lymphoepithelioma
* Locally advanced disease (stage III or IV [M0] disease)
* At least 1 unidimensionally measurable index lesion

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Bilirubin ≤ 1.5 times the upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3.0 times ULN
* AST and ALT ≤ 3.0 times ULN
* Creatinine ≤ 1.5 times ULN
* No concurrent serious systemic disorder that, in the opinion of investigator, would compromise the patient's ability to complete the study
* No serious cardiac condition, including any of the following:

  * Myocardial infarction within the past 6 months
  * Angina
  * NYHA class III-IV heart disease
* No active infection requiring IV antibiotics, including active tuberculosis or HIV
* No other malignancy within the past 5 years except basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* Able to comply with protocol or study procedures

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (complete or partial response) as assessed by RECIST criteria

SECONDARY OUTCOMES:
Progression-free survival
Overall survival
Toxicity as assessed by NCI CTCAE v3.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hang Kim, MD, Study Chair — Yonsei University
Locations (1):
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea